CLINICAL TRIAL: NCT01166295
Title: Development of a Bedside Pain Assessment Kit for Postherpetic Neuralgia
Acronym: BSTK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Analgesic Solutions (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Nathaniel Katz, MD,MS - Principal Investigator, Analgesic Solutions
Other Study IDs: MRK.008a.2010
Record Dates: First submitted 2010-07-12; First posted 2010-07-21 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-08

CONDITIONS: Neuralgia; Herpes Zoster
MeSH Terms: conditions — Neuralgia; Herpes Zoster

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Post herpetic neuralgia (PHN) is an undertreated condition. It is a type of neuropathic pain (NP), or pain caused by abnormal activity of sensory nerves. Its mechanisms are not fully understood, and medication trials for PHN pain and other types of NP are frequently unsuccessful.

There has been extensive investigation aimed at identifying and understanding the specific mechanisms of NP. While some of these tests are inexpensive and easy to perform at the bedside, many require expensive tools and highly equipped laboratory facilities. Further, there is no standard method for assessment of pain in NP patients.

The investigators aim to test a Bedside Sensory Testing Kit (assessment for Neuropathic Pain) on a small number of patients with PHN.

The purpose of the Kit is to identify mechanisms of pain. The goal of this research is to design a way to classify patients with PHN based on what mechanisms are causing their pain, since this may help predict the best medications for individual patients.

DETAILED DESCRIPTION:
We hypothesize: (a) that a Bedside Sensory Testing Kit for PHN can be designed such that it works efficiently with Subjects and Investigators, is tolerated well by Subjects, and is statistically reliable between Investigators; (b) that the sensory testing kit can distinguish between PHN patients with different sensory qualities to their pain which may be caused by different underlying pain mechanisms.

The subjects will be patients with postherpetic neuralgia who voluntarily participate and meet eligibility criteria. The study participants will complete a brief questionnaire and undergo three rounds of the BSTK, performed by two study investigators. The items in the BSTK correspond to a series of sensory assessments, each of which are aimed to contribute to the characterization of individuals' PHN pain.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 40 and 85 years old.
* Physician documentation of history of postherpetic neuralgia must be provided; pain persisting more than 3 months/90 days after a patient's vesicular rash (shingles) has healed.
* Subject is able to speak, read and write in English and comply with all study procedures;
* Subject is willing to voluntarily sign and date an Informed Consent Form, approved by an IRB, prior to the conduct of any study-specific procedures;
* Subject must be willing to abstain from PRN (as needed) pain medicine for 12 hours prior to the study but may continue their standing doses of pain medicine.

Exclusion Criteria:

* Subject is pregnant and/or breast-feeding.
* Subjects with additional sources of chronic pain will not be allowed if the severity of pain in additional locations is severe enough to compromise assessment of PHN pain. This will be left to the Investigator's discretion.
* Subject has a medical condition, other than PHN, that is not well-controlled with treatment; or the subject has any clinically significant condition that would, in the opinion of the investigator, preclude study participation, interfere with the assessment of pain, or pose unacceptable risk to the participant.
* Subject has been enrolled in another study within 30 days.
* Subject has a known contact allergy to surgical skin markers.
* In the judgment of the investigator, the subject has a psychiatric or psychological disorder that would interfere with the completion of the study, confound the study results, or pose patient risk.
* Subject has neuropathy or nerve fiber disease other than PHN (e.g., diabetic peripheral neuropathy).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample patients with postherpetic neuralgia who voluntarily participate and meet eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-10 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Demonstrate usability of the BSTK. | Subject Duration in the study is one (1) clinic visit ( approximatley 2-3 hours). We expect 10 weeks of open enrollment. Total study timeline is 4 months(1 month start up, 2 months enrollment, 1 month clean and analysis, 2 weeks final CSR.
  Analysis of subject feedback regarding clarity of instructions, burden of study procedures, and overall experience.
  Analysis of investigator observations regarding clinical feasibility, investigator burden, and overall experience.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Katz, MD, MS, Principal Investigator — Analgesic Solutions
Locations (1):
- Analgesic Solutions, Natick, Massachusetts, United States